Single-center, Prospective, Non-Randomized

Control Clinical Trial of Retro - auricular Single - site

Endoscopic Versus Open Surgery in Patients with

Early Stage Papillary Thyroid Carcinoma

Study Protocol

Version date: January, 19, 2022

| | Single center Prognective Non Bandamized Central Clinical Trial of |
|---|---|
| Official Title | Single-center, Prospective, Non-Randomized Control Clinical Trial of |
| Official Title | Retro - auricular Single - site Endoscopic Versus Open Surgery in |
| | Patients with Early Stage Papillary Thyroid Carcinoma The goal of this pap randomized control clinical research study is to |
| Brief | The goal of this non randomized control clinical research study is to |
| | compare the cosmetic outcomes and efficiacy of retro - auricular single - |
| Summary | site endoscopic thyroid lobectomy and central lymph node dissection |
| 0 1111 | against conventional resection. |
| Conditions | Age: 18~70 years.Patients with early stage papillary thyroid carcinoma. |
| | Primary Outcome Measure: postoperative cosmetic satisfaction |
| | scores |
| | Secondary Outcome Measures: |
| Outcome | Cosmetic outcome: postoperative Vancouver Scar Scale |
| Measures | Surgical outcomes: CRP level, SAA level, intraoperative blood |
| | loss, VAS pain score, Operative time. |
| | Clinicopathologic characteristics: tumor size, number of lymph |
| | nodes, the positive rate of lymph nodes. |
| | Complication: complication rates and types |
| | RASSET group |
| Study | early stage papillary 1:1 N=40 Postoperative cosmetic |
| Process | Non-Randomized Open group satisfaction scores |
| | N=40 |
| Sample | 80(40 VS 40) |
| Size | , , , |
| | Age 18-70 years old, no gender restrictions. |
| | Fine-needle aspiration cytology(FNA) confirmed papillary thyroid |
| | carcinoma(PTC). |
| Inclusion | Early stage PTC (stage T1N0M0). |
| Criteria | Preoperative ultrasonography showed unilateral glandular lobe |
| | malignant tumor and the largest diameter was not more than 2cm, |
| | without cervical lymph node metastasis and extensive metastasis. |
| | Patients undergoing thyroid lobectomy and central lymph node |
| | dissection. |
| | Patients who have signed an approved Informed Consent. |
| | Patients who do not accept case data collection for various reasons. |
| Exclusion | The clinical data unfit this study (at the discretion of the investigator). Deticate the base of the second state of |
| Criteria | Patients who have undergone neck surgery or radiotherapy before this |
| | trail. |
| | Patients who have uncontrolled hyperthyroidism. |
| Elimination | Patients who violated the requirements of the research protocol. |
| Criteria | The quality of data records is incomplete and inaccurate. |
| | Lost cases. |
| Study<br>Completion | 2023-06-30 |
| Locations | 1 |
| Locations | ' |

| Groups | RASSET group VS traditional open thyroid lobectomy group |
|---|---|
| Masking<br>and<br>Allocation | None (Open Label). Non-Randomized(patient decided his surgery approach). |
| Statistical<br>Analysis<br>Plan | In this clinical study, the test level $\alpha$ was set to be 0.05 on both sides; the test efficiency Power (ie, 1- $\beta$ ) was selected as 0.8 (ie, type II error $\beta$ =0.2); The sum standard deviation is 5.54 $\pm$ 1.75, and the mean and standard deviation of the score of the cosmetic effect evaluation scale of the experimental group is expected to be 3.92 $\pm$ 1.4 1. The 1:1 parallel control method is used, and the sample size calculation formula is based on the mean comparison of the two samples. According to the calculation of PASS software, this study requires a sample size of about 72 people (36 cases in each group). Considering the 10% dropout rate, the required sample size for each group is 40 cases, and a total of 80 cases in the two groups are required. All analyses were performed using SPSS 26.0, and a $P$ value less than 0.05 was considered significant. Normally distributed quantitative data are represented by mean (SD) [range]. Non-normally distributed quantitative data are represented by $M$ ( $Q_R$ ). Comparison between groups was performed using the Mann-Whitney U test. Categorical data are expressed as frequencies and percentages. Comparisons between groups were performed using the $\chi^2$ test or Fisher's exact test. |

# Study Protocol

## 1.Background

Thyroid cancer is one of the most common malignant tumors in the head and neck. Among it, papillary thyroid carcinoma accounts for about 70% of thyroid cancer. The degree of malignancy is low, but there is a tendency for multicentricity, and cervical lymph node metastasis occurs early. Due to the development of diagnosis technology, the amount of papillary microcarcinoma is getting higher and higher. At the same time, the change of aesthetic makes young women pursue a scarless neck<sup>1, 2</sup>. Surgery is the first choice of treatments for early-stage thyroid cancer.<sup>3, 4</sup> Traditional open surgery tended to leave a long scar on the neck, which affects the cosmetic outcome. At present, many reported approaches, such as trans-areola approach<sup>5</sup>, trans-axillary approach<sup>6</sup>, trans-oral approach <sup>7, 8</sup>or some combined approaches<sup>9</sup>, all have wider flap dissection or greater body trauma, and at the same time, these above approaches are difficult to achieve complete dissection of central lymph nodes<sup>10</sup>.

Therefore, based on the experience of transauricular hairline endoscopic thyroidectomy<sup>11-13</sup>, we established a new operative method-the Retro-auricular single-site endoscopic thyroidectomy (RASSET). The incision is only 3cm and located at the

posterior sulcus of the auricle, which can meet the cosmetic needs. Compared with other endoscopic approaches, the dissection area is small and the flap dissection is small, which may reduce the surgical trauma. The RASSET is easy to resect the upper pole of the thyroid gland, and can achieve complete dissection of the central lymph nodes. The article titled "A comparative study between retro - auricular single - site endoscopic thyroidectomy and transoral endoscopic thyroidectomy vestibular approach: a single - center retrospective analysis " has been published in " Chin J Surg "<sup>14</sup>. Guangdong Medical Information Research Institute recognized that there was no report of endoscopic thyroid surgery for this approach at home and abroad, and it also passed the new technology evaluation in the Sun Yat-sen University Cancer Center, and was recognized as an international leader.



**Figure 1.** A:Sun Yat-sen University Cancer Center Certificates(international innovation). **B**:Guangdong Medical Information Research Institute Certificates(no report of this approach). **C**:Zhonghua Wai Ke Za Zhi(a new approach).

## 2. Study purpose

#### Primary purpose:

Comparing the cosmetic outcomes of the retroauricular approach and the open group by comparing postoperative cosmetic satisfaction scores. (Appendix 1)

- Secondary purpose:
  - Comparing the degree of surgical trauma between the retroauricular group and the open group by comparing the level of CRP and SAA, blood loss, VAS pain score, and postoperative drainage.
  - Comparing the clinicopathologic characteristics between the retroauricular group and the open group by comparing the number of resected lymph nodes, and the positive rate of lymph nodes.
  - > Comparing the safety between the retroauricular group and the open group by comparing the types and rate of complications between the two groups.
- Primary Outcome Measure: postoperative cosmetic satisfaction scores
- Secondary Outcome Measures:
  - Cosmetic outcome: postoperative Vancouver Scar Scale

- > Surgical outcomes: CRP level, SAA level, blood loss, VAS pain score, postoperative drainage volume, Operative time.
- ➤ Clinicopathologic characteristics: tumor size, number of lymph nodes, the positive rate of lymph nodes.
- Complication: complication rates and types.



Figure 2. Kyung Tae's authorization

## 3. Study Eligibility

- Inclusion Criteria:
  - > Age 18-70 years old, no gender restrictions.
  - Fine-needle aspiration cytology(FNA) confirmed papillary thyroid carcinoma(PTC).
  - > Early stage PTC (stage T1N0M0).
  - Preoperative ultrasonography showed unilateral glandular lobe malignant tumor and the largest diameter was not more than 2cm, without cervical lymph node metastasis and extensive metastasis.
  - Patients undergoing thyroid lobectomy and central lymph node dissection.
  - Patients who have signed an approved Informed Consent.
- Exclusion Criteria:

- > Patients who do not accept case data collection for various reasons.
- > The clinical data unfit this study (at the discretion of the investigator).
- > Patients who have undergone neck surgery or radiotherapy before this trail.
- Patients who have uncontrolled hyperthyroidism.

#### Withdrawal criteria:

(A withdrawal case refers to a patient who withdraws from treatment for various reasons in study. Patients with the following conditions will be withdrawn from investigational treatment.)

- The patient himself or his legal representative requests to withdraw.
- In the opinion of the investigator, the patient's continued participation in the study will be detrimental to his health.

#### • Elimination Criteria:

- > Patients who violated the requirements of the research protocol.
- The quality of data records is incomplete and inaccurate.
- Lost cases.

## 4. Case Screening

#### examination items

All cases must complete the following examination items before being considered for entry into this study. It is generally required to be completed within 7 days before treatment.

- > Complete medical history and comprehensive physical examination, including symptoms, signs and specialist examination.
- Check items that must be done before routine treatment, including:Blood routine: neutrophil/lymphocyte ratio,Coagulation function: d-dimer,Serological tests: CRP, SAA, procalcitonin, calcium level,Thyroid function: TSH level, parathyroid hormone level,Thyroid ultrasonography, thyroid Computed tomography scan if necessary,Chest X-ray, abdominal ultrasonography, electrocardiogram.

# The above examinations are all routine preoperative examinations, which do not cause additional financial burden on patients.

## Case screening

According to various examinations, those who meet the inclusion criterias are screened out. The patients entered the study after completing the required examinations and being evaluated according to the inclusion criterias. Then sign the informed consent form and get treatment.

# 5. Study Process

Figure 3. flowchart



## Surgical Technique

Retro-auricular single-site endoscopic thyroidectomy (RASSET)

For the RASSET technique, in the beginnig, patient was placed in a supine position with slight neck bending. When the lower pole of the thyroid gland was going to be dissected, the patient was placed in a supine position with slight neck extension. Mark the operation path on the surface. Slit the skin, subcutaneous tissue and superficial cervical fascia in turn. Expose the middle branch of the great auricular nerve and the sternocleidomastoid muscle under direct vision. The working space was created in the superficial layer of deep cervical fascia between the sternocleidomastoid muscle and the platysma muscle, which meets the principle of membrane anatomy. The area of flap dissection just includes the anterior cervical muscle and the anterior edge of the sternocleidomastoid muscle, which is so narrow to minimize the traumatic dissection. Pulling apart the anterior cervical muscle and the sternocleidomastoid muscle along the deep cervical fascia can fully expose the thyroid gland, the recurrent laryngeal nerve (RLN) and common carotid artery that are surrounded by the middle layer of deep cervical fascia and ensure that tumor and central lymph nodes en - bloc resection can be operated in the middle layer of deep cervical fascia to conform the natural anatomical region. For details, please refer to "A comparative study between retro - auricular single - site endoscopic thyroidectomy and transoral endoscopic thyroidectomy vestibular approach: a single - center retrospective analysis".



Figure 4. model and practical operation

## traditional open surgery

For traditional open surgery, the patient was placed in a supine position. A 4-6cm transverse incision was made. Subplatysmal flaps were dissected up to the thyroid cartilage and down to the sternal notch. The strap muscles were separated in the midline to expose the thyroid gland. Lateral dissection of the thyroid gland was performed. The middle thyroid vein was ligated. Superior thyroid vessels were individually ligated close to the thyroid gland. The RLN was identified and dissected near the inferior thyroid artery. Branches of the inferior thyroid vessels were ligated, preserving the lower parathyroid gland. Berry ligament was then dissected, and finally the isthmus was transected. The thyroid and central lymph nodes were resected. For details, please see "Clinical Practice and Skills in Head and Neck Oncology Surgery".

#### 7. Outcome Measures

Baseline Characteristics of Patients

Gender, Age, BMI, Tumor size, Pathological type, Tumor location, ASA grade.

- Postoperative Outcomes
  - ➤ Cosmetic outcome: postoperative Vancouver Scar Scale 1 and 3 months from surgery, postoperative cosmetic satisfaction scores 1 month from surgery.
  - > Surgical outcomes: CRP level, SAA level, Drainage volume (ml), intraoperative blood loss, VAS pain score, Operative time.
  - ➤ Clinicopathologic characteristics: tumor size, number of lymph nodes, the positive rate of lymph nodes.
  - Complications: complication rates and types.
- Primary Outcome Measure: postoperative cosmetic satisfaction scores 3months from surgery.

## 8. Code of Ethics

#### Informed consent

Before each patient was enrolled in this study, the research investigators are responsible for a complete and comprehensive introduction to the surgical method of this study, its possible side effects and possible risks, and let patients know their rights, risks and benefits to be assumed. Patients should have signed informed consent before enrollment.

Ethical norms and policies and regulations

This clinical trial must comply with the Declaration of Helsinki (2000 Edition), the Good Clinical Practice (GCP) promulgated by the SFDA, and related regulations. Before the start of the trial, the study could be started only after the protocol was approved by the ethics committee of the lead unit. Any modification of the trial protocol during clinical research should be reported to the ethics committee and filed.

Obtaining ethics approval

Ethical approval has been obtained.

## 9. Quality Assurance

In order to ensure that this trial can be carried out in strict accordance with the clinical research protocol, during the entire process of the clinical trial, clinical investigators and clinical sponsors should behave in strict accordance with the requirements of the Good Clinical Practice for Drugs (GCP), and be sure to follow the trial procedures. Standardized, accurate test data, and reliable research conclusions. Specific requirements are as follows:

- Requirements for collaborators:
  - ➤ Lectures on clinical programs, CRF filling, etc. are given to the researchers before the clinical start.
  - > Send clinical monitors to conduct on-site inspections.
  - Ensure that the researchers can keep in touch with the researchers at any time by telephone or email.
- Requirements for researchers:
  - Responsible for obtaining the "Informed Consent" signed by each subject or his agent.
  - Complete the case report form (CRF) carefully as required.
  - Regular visits.
  - > Completely maintain records of clinical records, and original medical records of subjects.

## 10. Data Processing and Preservation

#### Case report form (CRF)

The case report form should be filled out by investigators, and the CRF form should be filled out in time to ensure accurate content and timely summary. Generally, the CRF form should not be altered. If there is an error that needs to be revised, it should be signed at the revised place. The CRF form is in triplicate, and after the trial is over, it will be handed over to the clinical team leader hospital, the sponsor and the trial hospital for preservation. Data entry was performed after the completed case report was reviewed by the clinical monitor. The contents of the case report form are no longer modified.

#### Create a database

After receiving the CRF form, the statistician will verify the question by the researcher, and the researcher should answer and return as soon as possible. Statisticians will establish a database at the same time. After the database is reviewed, the data will be locked by the principal investigators, sponsors, statistician and clinical monitors. To ensure data security, irrelevant personnel cannot access and modify the data, and the data must be backed up.

### Storage of data

The researcher should keep the data intact. According to the principle of GCP in China, for the investigators or hostipals, the data storage should be more than 5 years.

## 11. Statistical analysis

Professional statisticians undertake statistical analysis tasks and participate in the whole process from experimental design, implementation to analysis and summary. After the study protocol and case report form are completed, a statistical analysis plan shall be formulated. After some necessary modifications shall be made during the study process as required, and a statistical analysis report shall be provided after the data analysis is completed.

### Sample size

In this clinical study, the test level  $\alpha$  was set to be 0.05 on both sides. the test efficiency Power (ie, 1- $\beta$ ) was selected as 0.8 (ie, type II error  $\beta$ =0.2). The sum standard deviation is 5.54 $\pm$ 1.75, and the mean and standard deviation of the score of the cosmetic effect evaluation scale of the experimental group is expected to be 3.92 $\pm$ 1.41. The 1:1 parallel control method is used, and the sample size calculation formula is based on the mean comparison of the two samples. According to the calculation of PASS software, this study requires a sample size of about 72 people (36 cases in each group). Considering the 10% dropout rate, the required sample size for each group is 40 cases, and a total of 80 cases in the two groups are required.

#### Statistical Analysis

All analyses were performed using SPSS 26.0, and a P value less than 0.05 was considered significant. Normally distributed quantitative data are represented by mean (SD) [range]. Non-normally distributed quantitative data are represented by M (QR). Comparison between groups was performed using the Mann-Whitney U test. Categorical data are expressed as frequencies and percentages. Comparisons between groups were performed using the \( \text{2} \) test or Fisher's exact test.

## 12. Follow-up

During the study period, each enrolled case was independently archived and registered for evaluation (CRF), and a resident physician was to be hired to be responsible for follow-up, registration, filling, and storage. After the end of treatment, the enrolled patients will be reviewed in the outpatient clinic in the first month after surgery, and then will be followed up regularly for 3-6 months until the death of the patient or the end of the study. The content of each review must include: thyroid function, parathyroid hormone level, thyroid ultrasonography. Questionnaires were conducted in the first and third months after surgery, and the scores of the Beauty Evaluation Scale and the Postoperative Scar Scale

were recorded and counted.

## 13. Study Start and Completion

Study Start: March 1, 2022

Anticipated Study Completion: June 30, 2023

A total of 40 patients in the RASSET group and 40 patients in the open group will be Enrolled, follow up 1 and 3 months after the operation, and the clinical data will be collected and analyzed statistically.

# **References:**

- **1.** Anuwong A, Ketwong K, Jitpratoom P, Sasanakietkul T, Duh Q. Safety and Outcomes of the Transoral Endoscopic Thyroidectomy Vestibular Approach. *Jama Surg.* 2018;153(1):21.
- **2.** Lee DW, Ko SH, Song CM, Ji YB, Kim JK, Tae K. Comparison of postoperative cosmesis in transaxillary, postauricular facelift, and conventional transcervical thyroidectomy. *Surgical Endoscopy*. 2020;34(8):3388-3397.
- **3.** Filetti S, Durante C, Hartl D, et al. Thyroid cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. *Ann Oncol.* 2019;30(12):1856-1883.
- **4.** Haugen BR, Alexander EK, Bible KC, et al. 2015 American Thyroid Association Management Guidelines for Adult Patients with Thyroid Nodules and Differentiated Thyroid Cancer: The American Thyroid Association Guidelines Task Force on Thyroid Nodules and Differentiated Thyroid Cancer. *Thyroid*. 2016;26(1):1-133.
- **5.** Liang J, Zhan L, Xuan M, et al. Thyroidectomy for thyroid cancer via transareola single-site endoscopic approach: results of a case-match study with large-scale population. *Surgical Endoscopy*. 2021.
- **6.** Alramadhan M, Choe JH, Lee JH, Kim JH, Kim JS. Propensity score-matched analysis of the endoscopic bilateral axillo-breast approach (BABA) versus conventional open thyroidectomy in patients with benign or intermediate fine-needle aspiration cytology results, a retrospective study. *Int J Surg.* 2017;48:9-15.
- 7. Nguyen HX, Nguyen HV, Nguyen LT, Nguyen TTP, Le QV. Transoral Endoscopic Thyroidectomy by Vestibular Approach with Central Lymph Node Dissection for Thyroid Microcarcinoma. *J Laparoendosc Adv S.* 2021;31(4):410-415.
- **8.** Nakajo A, Arima H, Hirata M, et al. Trans-Oral Video-Assisted Neck Surgery (TOVANS). A new transoral technique of endoscopic thyroidectomy with gasless premandible approach. *Surgical Endoscopy*. 2013;27(4):1105-1110.
- **9.** Berber E, Bernet V, Fahey TR, et al. American Thyroid Association Statement on Remote-Access Thyroid Surgery. *Thyroid*. 2016;26(3):331-337.
- **10.** Duek I, Duek OS, Fliss DM. Minimally Invasive Approaches for Thyroid Surgery—Pitfalls and Promises. *Curr Oncol Rep.* 2020;22(8).
- **11.** Schardey HM, Barone M, Portl S, von Ahnen M, von Ahnen T, Schopf S. Invisible scar endoscopic dorsal approach thyroidectomy: a clinical feasibility study. *World J Surg*. 2010;34(12):2997-3006.
- **12.** Schardey HM, Schopf S, Kammal M, et al. Invisible scar endoscopic thyroidectomy by the dorsal approach: experimental development of a new technique with human cadavers and preliminary clinical

results. Surg Endosc. 2008;22(4):813-820.

- **13.** Chung E, Park M, Cho J, et al. A Prospective 1-Year Comparative Study of Endoscopic Thyroidectomy Via a Retroauricular Approach Versus Conventional Open Thyroidectomy at a Single Institution. *Ann Surg Oncol.* 2015;22(9):3014-3021.
- **14.** Dong F, Ao Y, Li MT, et al. [A comparative study between retro-auricular single-site endoscopic thyroidectomy and transoral endoscopic thyroidectomy vestibular approach: a single-center retrospective analysis]. *Zhonghua Wai Ke Za Zhi.* 2021;59:891-896.

# **Appendix**

## Appendix 1 Cosmetic satisfaction questionnaire

Q1. How satisfied are you with your neck scar or a scarless neck?

Very satisfied(1) Satisfied(2) Average(3) Dissatisfied(4) Verydissatisfied(5)

Q2. How satisfied are you with the contour of your neck?

Very satisfied(1) Satisfied(2) Average(3) Dissatisfied(4) Verydissatisfied(5)

Q3. Do you think others look at your neck scar?

Absent (0) Sometimes (1) Frequent (2) Always (3)

Q4. Do you try to conceal your scar?

Absent (0) Sometimes (1) Frequent (2) Always (3)

Q5. Does your neck scar influence your choice of clothes?

Absent (0) Sometimes (1) Frequent (2) Always (3)

Q6. How often do you think about your scar?

Absent (0) Sometimes (1) Frequent (2) Always (3)

# Appendix 2 Vancouver scar scale score

| | Feature | Score |
|---|---|---|
| Vascularity | Normal<br>Pink<br>Red<br>Purple | 0<br>1<br>2<br>3 |
| Pigmenta-<br>tion | Normal Hypo-pigmentation Mixed-pigmentation Hyper-pigmentation | 0<br>1<br>2<br>3 |
| Pliability<br>(Elasticity) | Normal Supple (flexible with minimal resistance) Yielding (giving way to pressure) Firm (inflexible, not easily moved, resistant to manual pressure) Banding (rope-like tissue that blanches with extension of the scar) Contracture (permanent shortening of scar, producing deformity or distortion) | 0<br>1<br>2<br>3<br>4<br>5 |
| Height | Flat < 2 mm 2-5 mm > 5 mm | 0<br>1<br>2<br>3 |
| Pain | None<br>Occasional<br>Requires medication | 0<br>1<br>2 |
| Itchiness | None<br>Occasional<br>Requires medication | 0<br>1<br>2 |

Appendix 3 AJCC 8th Edition/TNM Classification System for

Differentiated Thyroid Carcinoma

| | Stag | jing flowcha | art for differentiated thyroic | l cancer (AJC0 | 8e) | |
|---|---|---|---|---|---|---|
| Age<br>at diagnosis | M<br>category | Gross<br>ETE | Structures involved | Tumor<br>size | N<br>category | Stage |
| <55 years | MO<br>M1 | yes or no<br>yes or no | | any<br>any | any<br>any | <br> |
| ≥ 55 years | МО | no | | ≤ 4 cm (T1-2)<br>> 4 cm (T3a) | N0/Nx<br>N1a/N1b<br>any | <br> <br> |
| | | yes | only strap muscle (T3b)<br>s/cutaneous, larynx, trachea,<br>esophagus, RL nerve (T4a) | any | any<br>any | II<br>III |
| | | | prevertebral fascia,<br>encasing major vessels (T4b) | any | any | IVA |
| | M1 | yes or no | any or none | any | any | IVB |

| | TNM definitions (AJCC 8e) |
|---|---|
| for papil | lary, follicular, poorly differentiated, Hürthle cell, medullary, and anaplastic thyroid carcinomas |
| TX | Primary tumor cannot be assessed |
| T0 | No evidence of primary tumor |
| T1 | Tumor ≤ 2 cm in greatest dimension limited to the thyroid |
| T1a | Tumor ≤ 1 cm in greatest dimension limited to the thyroid |
| T1b | Tumor > 1 cm but ≤ 2 cm in greatest dimension limited to the thyroid |
| T2<br>T3* | Tumor > 2 cm but ≤ 4 cm in greatest dimension limited to the thyroid |
| | Tumor > 4 cm limited to the thyroid or gross extrathyroidal extension invading only strap muscles |
| T3a* | Tumor > 4 cm limited to the thyroid |
| T3b* | Gross extrathyroidal extension invading only strap muscles (sternohyoid) from a tumor of any size |
| T4 | Includes gross extrathyroidal extension into major neck structures |
| T4a | Gross extrathyroidal extension invading subcutaneous soft tissues, larynx, trachea, esophagus, |
| T 41- | or recurrent laryngeal nerve from a tumor of any size |
| T4b | Gross extrathyroidal extension invading prevertebral fascia or encasing carotid artery |
| NX | or mediastinal vessels from a tumor of any size Regional lymph nodes cannot be assessed |
| NO | No evidence of regional lymph nodes metastasis |
| N0a* | One or more cytologic or histologically confirmed benign lymph node |
| N0b* | No radiologic or clinical evidence of locoregional lymph node metastasis |
| N1* | Metastasis to regional nodes |
| N1a* | Metastasis to level VI or VII (pretracheal, paratracheal, or prelaryngeal/Delphian, or upper |
| ,,,, | mediastinal) lymph nodes; this can be unilateral or bilateral disease |
| N1b* | Metastasis to unilateral, bilateral, or contralateral lateral neck lymph nodes (levels I, II, III, IV, or V |
| | or retropharyngeal lymph nodes |
| MO | No distant metastasis |
| M1 | Distant metastasis |